CLINICAL TRIAL: NCT04719663
Title: The Modulatory Role of Communicated Treatment Rationale on Treatment Expectation Effects in Depression.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Psychotherapie-Ambulanz Marburg e.V. (Other)
Responsible Party: Principal Investigator, Winfried Rief, Prof. Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CRC 289 Project A16
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Condition: Major Depressive Disorder (MDD)
Keywords: Placebo effect; Treatment rationale; Depression; Expectations
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be blinded to the congruency condition. Outcome assessors (diagnosticians) will be blinded to treatment allocation and the congruency condition (both at the pre-measurement and at the post-measurement). The clinicians (care providers) who deliver the illness explanation and treatment rationale will be blinded to the participants' treatment allocation up to the point at which the respective treatment is delivered. This means that the clinician provides the treatment rationale (biological / psychological) without knowledge of whether a congruent or incongruent treatment will be delivered afterwards. The staff members who deliver the treatment (care providers) will be different to the clinician who delivers the rationales. Thus the treatment will be delivered without knowledge of whether a congruent or incongruent illness explanation was given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1. Congruent Rationale & Treatment: Biological/Pharmacol. (Experimental): Participants receive a biological illness explanation and treatment rationale. During treatment they receive a placebo pill (Buscopan).
  Interventions: Behavioral: Biological illness and treatment rationale; Drug: Active pharmacological placebo
- 2. Incongruent Rationale & Treatment: Psychological/Pharmacol. (Experimental): Participants receive a psychological illness explanation and treatment rationale. During treatment they receive a placebo pill (Buscopan).
  Interventions: Behavioral: Psychological illness and treatment rationale; Drug: Active pharmacological placebo
- 3. Congruent Rationale & Treatment: Psychological/Psychol. (Experimental): Participants receive a psychological illness explanation and treatment rationale. During treatment they receive a placebo psychological treatment (emotional writing).
  Interventions: Behavioral: Psychological illness and treatment rationale; Behavioral: Active psychological placebo
- 4. Incongruent Rationale & Treatment: Biological/Psychol. (Experimental): Participants receive a biological illness explanation and treatment rationale. During treatment they receive a placebo psychological treatment (emotional writing).
  Interventions: Behavioral: Biological illness and treatment rationale; Behavioral: Active psychological placebo
- 5. Natural course control (No Intervention): Participants receive no intervention and remain on the psychotherapy waiting list. Participants who are recruited externally and are not on a waiting list, will be offered the option to join the waiting list.

INTERVENTIONS:
Behavioral: Biological illness and treatment rationale — Depression is described as a brain disorder and the role of monoamine, brain structures, and brain functions are reported as central mechanisms of relevance for its etiology and treatment. Biological processes are illustrated using typical charts and visualizations. Psychological influences are mentioned, but only as a byproduct of the disorder.
  Arms: 1. Congruent Rationale & Treatment: Biological/Pharmacol.; 4. Incongruent Rationale & Treatment: Biological/Psychol.
Behavioral: Psychological illness and treatment rationale — Depression is described as a psychological disorder resulting from emotion regulation deficits. The suppression of emotions receives a special role in explaining depression. The psychological processes are illustrated using charts and visualizations. Biological aspects are mentioned, but only as a byproduct of the disorder.
  Arms: 2. Incongruent Rationale & Treatment: Psychological/Pharmacol.; 3. Congruent Rationale & Treatment: Psychological/Psychol.
Drug: Active pharmacological placebo — The active placebo pill does not have direct effects on the brain. Buscopan (butylscopolamine, 10 mg daily, 1 pill in the morning) does not cross the blood-brain barrier, yet induces some smaller side effects that resemble those of antidepressants (e.g., mouth dryness, fatigue, nausea). Treatment duration is 4 weeks. The rationale is briefly explained to participants as "stimulating the biological balance in humans with depression, using a well-tolerated drug similar to Buscopan, which is well-known from pain treatments.
  Arms: 1. Congruent Rationale & Treatment: Biological/Pharmacol.; 2. Incongruent Rationale & Treatment: Psychological/Pharmacol.
Behavioral: Active psychological placebo — "Emotional writing" consists of writing about emotional experiences (4 sessions, one per week, 30 minutes each). The study instructor will be present displaying standard psychotherapeutic attitudes but will not read the participant's notes. The rationale for this treatment is briefly explained as "improving the dealing" with emotions to achieve a psychological balance in humans with depression.
  Arms: 3. Congruent Rationale & Treatment: Psychological/Psychol.; 4. Incongruent Rationale & Treatment: Biological/Psychol.

SUMMARY:
Placebo groups in clinical trials on depression show impressive improvements. Yet, there is little research on the mechanism underlying this effect. The aim of this study is to assess how patients' treatment expectations modulate the placebo treatment effects.

We expect that patients' treatment expectation determines placebo responses and treatment outcomes, and that this expectation is influenced by the disorder explanations (information about the illness models) typically provided during the initial medical encounters that precede treatment.

In the study we aim to manipulate depressed patients' expectations by providing two different clinician-delivered illness and treatment rationales (biological/ psychological). Patients will then receive placebo treatment (pharmacological/ psychological), that is either congruent or incongruent with the previously communicated treatment rationale.

Hypotheses:

1. Providing a treatment-congruent treatment rationale leads to a better outcome than providing treatment-incongruent rationales.
2. Treatment-congruent explanations reduce the risk of side effect development, in particular in the medication arm.
3. Inter-individual differences in the effect of provided treatment rationale are associated with pre-treatment experiences and expectations, depression severity and comorbid anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depression according to the 'Structured Clinical Interview for DSM-V' (SCID)
* Age>17
* Comorbidity is allowed if major depression is the dominant clinical problem
* Concordant medication is allowed if kept constant for the four weeks before and until the end of the trial (with the exception of benzodiazepines and if not contraindicated together with Buscopan)
* Fluency in German
* Informed consent

Exclusion Criteria:

* Severe depression (BDI> 30) or suicidality
* Psychosis
* Significant neurological diseases
* Other mental or physical disorder with substantial influence on disability
* Benzodiazepine intake
* Any intolerance against Buscopan and sucrose or any medical condition/treatment conflicting with Buscopan intake

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Change in depression severity scores after 4 weeks of treatment - 'Montgomery Asberg Depression Scale' (MADRS) | Baseline, post-treatment (4 weeks after start of treatment)
  Expert rating to assess depression severity; 10 items; each item is rated on a 7-point scale (0-6); total scores range between 0-60 (higher scores indicate more severe depression)

SECONDARY OUTCOMES:
Change in depressive symptom scores after 4 weeks of treatment- 'Beck Depression Inventory' (BDI-II) | Baseline, post-treatment (4 weeks after start of treatment), and at follow-up (1 week later)
  Self-report questionnaire to assess subjective depression symptomatology; 21 items (each item response is scored 0-3); total scores range from 0 - 63 (higher scores indicate more depressiveness)
Change in subjective disability scores after 4 weeks of treatment - adaptation of 'Pain Disability Index' (PDI) | Pre-treatment (2-7 days after baseline), post-treatment (4 weeks after start of treatment), and at follow-up (1 week later)
  Self-report questionnaire to assess illness burden; 7 items; each item rated on a 0 (no disability)-10(maximum disability) standardized numerical analogue scale; total scores range from 0-70 (higher scores indicate more disability)
Change in 'Generic Assessment of Side-Effects' scores (GASE) after 4 weeks of treatment | Pre-treatment (2-7 days after baseline), post-treatment (4 weeks after start of treatment), and at follow-up (1 week later)
  Self-report questionnaire to assess experience of side effects; 36 items; each item describes a side-effect symptom which is rated on a 4-point scale from 0 (not present)-3 (strong experience); total scores range from 0-108 (higher scores indicate stronger experience of side effects)
Change in treatment expectations at the start of treatment - 'Treatment Expectation Questionnaire' (TEX-Q) | Baseline, pre-treatment (2-7 days after baseline)
  Self-report questionnaire to assess expectations about treatment outcomes; 15 items; each rated on a 0 (no expectation of improvement)- 10(most improvement imaginable) numeric scale; total scores range from 0-150 (higher scores indicate better treatment expectations)
Change in subjective stress scores after 4 weeks of treatment - 'Perceived Stress Scale' (PSS-10) | pre-treatment (2-7 days after baseline), post-treatment (4 weeks after start of treatment), and at follow-up (1 week later)
  Self-report questionnaire to assess subjective stress experience; 10 items; each item is rated on a 5-point scale from 0(never) to 4(very often); total scores range between 0 and 40 (higher scores indicate more subjective stress)
Change in anxiety scores after 4 weeks of treatment - 'State-Trait-Anxiety- Depression-Inventory' (STADI) | State scale: Baseline; pre-treatment (2-7 days after baseline), post-treatment (4 weeks after start of treatment) and at follow-up (1 week later); Trait scale only measured at baseline
  Self-report questionnaire to assess state and trait anxiety and depression; 40 (20 state scale; 20 trait scale) items; each item is rated on a 4-point scale from 1(not at all) to 4(very much); total scores per scale range between 20 and 80 (higher scores indicate more anxiety)

OTHER OUTCOMES:
Treatment adherence | Once per week (during the 4-week treatment period)
  Count of remaining pills per week; participation in weekly therapy sessions
Common biological stress markers | Baseline
  Salivary Alpha-Amylase and cortisol levels
Current treatment effects after 4 weeks of treatment | post-treatment (4 weeks after start of treatment)
  Generic questions to assess perceived treatment effects; 3 items, each rated on a 0(no improvement) - 10(most improvement imaginable) numeric scale; total scores range from 0-30 (higher scores indicate better treatment expectations)
Current treatment effects at follow-up | at follow-up (1 week after end of treatment)
  Generic questions to assess perceived treatment effects; 3 items, each rated on a 0(no improvement) - 10(most improvement imaginable) numeric analogue scale; total scores range from 0-30 (higher scores indicate better treatment expectations)
Change in generic expectations about antidepressants at the start of treatment | Baseline; pre-treatment (2-7 days after baseline)
  Generic questions assess pre-existing expectations about antidepressants; 3 items; items are rated on a 0(no expectation of improvement) - 10(most improvement imaginable) numeric analogue scale; total scores range from 0-30 (higher scores indicate better antidepressant treatment expectations)
Change in generic expectations about psychotherapy at the start of treatment | Baseline, pre-treatment (2-7 days after baseline)
  Generic questions to assess pre-existing expectations about psychotherapy; 3 items; items are rated on a 0(no expectation of improvement) - 10(most improvement imaginable) numeric analogue scale; total scores range from 0-30 (higher scores indicate better psychotherapy treatment expectations)
'Somatosensory Amplification Scale' (SSAS) | Baseline
  Self-report questionnaire to assess amount of somatosensory amplification tendencies; 10 items; items are rated on a 5-point scale from 1(not at all true) - 5(extremely true); total scores range from 10-50 (higher scores indicate more somatosensory amplification)
'Behavioral Inhibition/Behavioral Approach System' Scale (BIS/BAS) | Baseline
  Self-report questionnaire to assess sensitivity to approach or avoidance goals; 24 items; each item is rated on a 4-point scale from 1(not at all true for me) to 4(very true for me)
Generic screening pre-experiences with antidepressants | Baseline
  Generic questions to assess pre-existing experiences with antidepressants; 4 items; if experience with antidepressants is indicated in item 1, the following 3 items are rated on a 0(no improvement) - 10(most improvement imaginable) numeric analogue scale; total scores range from 0-30 (higher scores indicate better past experiences with antidepressants)
Generic screening pre-experiences with psychotherapy | Baseline
  Generic questions to assess pre-existing experiences with psychotherapy; 4 items; if experience with psychotherapy is indicated in item 1, the following 3 items are rated on a 0 (no improvement)-10(most improvement imaginable) numeric analogue scale; total scores range from 0-30 (higher scores indicate better past experiences with psychotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Principal Investigator — Philipps University Marburg
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Philipps-University Marburg, Marburg, Germany

REFERENCES:
- [Derived] Henrich L, Wilhelm M, Lange P, Rief W. The role of the communicated treatment rationale on treatment outcome: study protocol for a randomized controlled trial. Trials. 2023 Aug 17;24(1):540. doi: 10.1186/s13063-023-07557-w. PMID 37592320